CLINICAL TRIAL: NCT00648466
Title: Single-Dose Fasting In Vivo Bioequivalence Study of Sumatriptan Succinate Tablets (100 mg; Mylan) to Imitrex® Tablets (100 mg; GlaxoSmithKline) in Healthy Volunteers
Brief Title: Fasting Study of Sumatriptan Succinate Tablets 100 mg to Imitrex® Tablets 100 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Wayne Talton, Mylan Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: SUMA-0358
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
MeSH Terms: interventions — Sumatriptan

ARMS (2):
- 1 (Experimental): Sumatriptan Succinate Tablets 100 mg
  Interventions: Drug: Sumatriptan Succinate Tablets 100 mg
- 2 (Active Comparator): Imitrex® Tablets 100 mg
  Interventions: Drug: Imitrex® Tablets 100 mg

INTERVENTIONS:
Drug: Sumatriptan Succinate Tablets 100 mg — 100mg, single dose fasting
  Arms: 1
Drug: Imitrex® Tablets 100 mg — 100mg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's sumatriptan succinate 100 mg tablets to GSK's Imitrex® 100 mg tablets following a single, oral 100 mg (1 x 100 mg) dose administration under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male and/or non-pregnant, non-lactating female.

   1. Women of childbearing potential must have negative serum beta human chorionic gonadotropin (beta-HCG) pregnancy tests performed within 14 days prior to the start of the study and on the evening prior to each dose administration. If dosing is scheduled on weekends, the HCG pregnancy test should be given within 48 hours prior to dosing of each study period. An additional serum (beta-HCG) pregnancy test will be performed upon completion of the study.
   2. Women of childbearing potential must practice abstinence or be using an acceptable form of contraception throughout the duration of the study. No hormonal contraceptives or hormone replacement therapy are permitted in this study. Acceptable forms of contraception include the following:

      1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      2. barrier methods containing or used in conjunction with a spermicidal agent, or
      3. surgical sterility (tubal ligation, oophorectomy or hysterectomy) or postmenopausal accompanied with a documented postmenopausal course of at least one year.
   3. During the course of the study, from study screen until study exit - including the washout period, women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive device. This advice should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women and all subjects within 15% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, hepatitis B and hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within the 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial dose of study medication.
   2. Use of any hormonal contraceptives and hormone replacement therapy within 3 months prior to study medication dosing.
   3. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to sumatriptan succinate or any other related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-11; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The 90% confidence interval for the LSMeans ratio of CPEAK, AUCL, and AUCI for the test and reference product should be between 80.00% and 125.00% for the natural log-transformed data. | Blood collections through 16 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Williams, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html